CLINICAL TRIAL: NCT04876846
Title: Trans-abdominal Fetal Pulse Oximetry; Tissue Light Scattering and Signal Integrity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raydiant Oximetry, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: GEN 3
Record Dates: First submitted 2021-04-27; First posted 2021-05-07 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Fetal Hypoxia
MeSH Terms: conditions — Fetal Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Interventional/Observational (Experimental): The Gen 3 device will be positioned on the maternal abdomen to measure light scattering and absorption for a period of about 10-20 minutes. A second measurement may be obtained for a total of up to 40 minutes. Subject's end their participation in the study after that time period.
  Interventions: Device: GEN 3 Monitoring of Fetus

INTERVENTIONS:
Device: GEN 3 Monitoring of Fetus — Measurement of tissue light scatter in the "body in body" during late term pregnancy and evaluation of signal integrity

SUMMARY:
The overall purpose of this study is to evaluate maternal-fetal tissue light scattering properties. The objectives of the study are: (i) integrate established mathematical principles of oxygen saturation to model with increasing accuracy the "body in a body" problem of fetus in mother; similar to existing pulse oximeters, the calculations will be integrated into software in the final commercial product; (ii) obtain human measurements against which both computational models and animal data can be compared.

DETAILED DESCRIPTION:
This is a prospective, observational, non-significant risk study. The study involves using non-invasive devices that measure fetal depth and tissue light scattering on the maternal abdomen. Ultrasound assessment will be performed, and multiple images taken at various locations on the abdomen. All images will be captured with minimal probe pressure applied to allow accurate ascertainment of depth. Images will be anonymized, and all study data will be coded with a unique identifier. Key maternal descriptive statistics will be recorded from the medical record including BMI, height, weight (kg), parity, age and gestational age.

The ISS device is a customized commercial frequency domain oximeter (Imagent, ISS Inc.; http://www.iss.com/biomedical/instruments/imagent.html) with multiple laser sources and multiple detectors. This instrument is safe, uses non-ionizing radiation.

The Raydiant Lumerah device is a non-invasive fetal pulse oximeter that measures fetal arterial oxygen saturation using safe, non-invasive, transabdominal near-infrared spectroscopy. The Lumerah device will be positioned on the maternal abdomen of women volunteers in the late 3rd trimester.

ELIGIBILITY:
Inclusion Criteria:

1. Women with singleton, healthy pregnancy at gestational age ≥ 36 weeks
2. Age > 18 years
3. Willing to come in for testing outside of routine business hours (including Saturdays)

Exclusion Criteria:

1. Age <18
2. Multiple gestation (twins, triplets)
3. Presentation other than vertex or breech
4. < 36 weeks of gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 9 (Actual)
Dates: Start 2021-04-24 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Fetal Signal | After 36 weeks of pregnancy
  Correlation of the fetal doppler signal with the ROSS device optional fetal signal.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rosen, MD, Study Director — Raydiant Oximetry
Locations (1):
- Yaron Friedman, MD, Inc., Walnut Creek, California, United States

IPD SHARING:
Plan to Share IPD: No
The data are specific to this device only.